CLINICAL TRIAL: NCT05906381
Title: A Clinical Trial of Dry Eye Symptom Mitigation by Oral Intake of Probiotics
Brief Title: Dry Eye Symptom Mitigation by Oral Intake of Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Nutrarex Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202300014B0
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2023-06

CONDITIONS: Dry Eye
Keywords: probiotics; dry eye; eye sore; eye strain
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Subjects will take a capsule of containing microcrystalline cellulose per day for 35 days.
  Interventions: Dietary Supplement: Placebo
- Treatment group (Experimental): Subjects will take a capsule of containing Streptococcus thermophilus per day for 35 days.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — A specific probiotics capsule product, containing Streptococcus thermophilus will be given to participants for oral intake for 35 days.
  Arms: Treatment group
Dietary Supplement: Placebo — A specific capsule product, containing microcrystalline cellulose will be given to participants for oral intake for 35 days.
  Arms: Control group

SUMMARY:
This study investigates whether the oral intake of a probiotics capsule product may relieve dry eye symptoms. Participants will be aged between 20 - 65 years of age, with confirmed diagnosis of dry eye status. The participants will be assessed for several parameters and asked to take 1 probiotics capsule per day for 35 days. The parameters will include ocular surface health, tear volume, tear quality, intraocular pressure, tear osmolarity and serum biochemical test. After the 35 days are completed, the participants will be assessed again for the same parameters.

DETAILED DESCRIPTION:
This investigation is a randomized, double-blind study. Subjects with confirmed diagnosis of dry eye are randomly assigned to control group or treatment group, and asked to orally intake 1 capsule of either placebo or probiotics per day. All participants will be assessed for parameters, including intraocular pressure, ocular surface health, tear film breakup time (TBUT), tear volume (Schirmer's test), tear osmolarity, ocular surface impression cytology, ocular surface disease index (OSDI) and serum biochemical tests for quantification of hyaluronic acid, sialic acid, glutathione contents.The assessments are conducted at day1 for baseline and after the 35-day oral intake. The parameters are used to compare and evaluate whether the probiotics can relieve dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 65 years
* with Schirmer's test results less than 10 mm or Ocular Surface Disease Index more than 25

Exclusion Criteria:

* evident ocular diseases such as cornea disease, cataract, vitreous degeneration, glaucoma, and retinopathy.
* diabetes
* hypertension
* or other chronic diseases or belong to vulnerable groups(pregnancy woman, prisoner, ethical minorities, economic or educationally disadvantaged subjects, disabled individuals such as those at terminal stage of tumorigenesis, blindness, terminal ill individuals)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Schirmer's Test Value from Baseline | on baseline and day36
  The Schirmer's Test is used to assess tear secretion volume. The amounts of tears are measured in total millimeters after 5 minutes has elapsed. Lower measurement amount is regarded as a parameter of presence of dry eye disease.
Change of Tear Film Breakup Time from Baseline | on baseline and day36
  Tear Break-Up Time is a measurement to reflect tear quality and is expressed in seconds. The shorter the Tear Break-Up Time, the poorer the tear film stability and quality. Lower measurement outcome (less than 10 seconds) is regarded as a parameter of presence of dry eye disease.
Ocular Surface Index Change from Baseline | on baseline and day36
  Ocular Surface Index is assessed with fluorescein staining to reflect ocular surface damages. The staining scale ranges from 0 to 3, from milder to severe status, where grade 0 shows no staining, and grade 3 shows extensive staining.
Tear Osmolality Change from Baseline | on baseline and day36
  Tear osmolality is used as a parameter of dry eye status.
Serum Biochemical Test | on baseline and day36
  To determine the effects of oral probiotics intake on the contents of hyaluronic acid, sialic acid, and glutathione in the serum.

SECONDARY OUTCOMES:
Ocular Surface Impression Cytology Change from Baseline | on baseline and day36
  To assess the status of conjunctival goblet cells and epithelium.
Ocular Surface Disease Index Score Change from Baseline | on baseline and day36
  A questionnaire is used to assess the health status on ocular surface, with higher scores indicating more severe status.
Intraocular Pressure Change from Baseline | on baseline and day36
  To determine the effects of intervention on intraocular pressure.

CONTACTS AND LOCATIONS:
Overall Officials: David Pei-Cheng Lin, Principal Investigator — Chung Shan Medical University
Locations (1):
- Jen-Ai Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrero-Vanrell R, Peral A. [International Dry Eye Workshop (DEWS). Update of the disease]. Arch Soc Esp Oftalmol. 2007 Dec;82(12):733-4. doi: 10.4321/s0365-66912007001200002. No abstract available. Spanish. PMID 18040913
- [Background] Fox RI, Chan R, Michelson JB, Belmont JB, Michelson PE. Beneficial effect of artificial tears made with autologous serum in patients with keratoconjunctivitis sicca. Arthritis Rheum. 1984 Apr;27(4):459-61. doi: 10.1002/art.1780270415. No abstract available. PMID 6712760
- [Background] Wilson WS, Duncan AJ, Jay JL. Effect of benzalkonium chloride on the stability of the precorneal tear film in rabbit and man. Br J Ophthalmol. 1975 Nov;59(11):667-9. doi: 10.1136/bjo.59.11.667. PMID 1203224
- [Background] Brito-Zeron P, Ramos-Casals M; EULAR-SS task force group. Advances in the understanding and treatment of systemic complications in Sjogren's syndrome. Curr Opin Rheumatol. 2014 Sep;26(5):520-7. doi: 10.1097/BOR.0000000000000096. PMID 25050925
- [Background] Sullivan DA, Krenzer KL, Sullivan BD, Tolls DB, Toda I, Dana MR. Does androgen insufficiency cause lacrimal gland inflammation and aqueous tear deficiency? Invest Ophthalmol Vis Sci. 1999 May;40(6):1261-5. PMID 10235562
- [Background] Schrader S, Mircheff AK, Geerling G. Animal models of dry eye. Dev Ophthalmol. 2008;41:298-312. doi: 10.1159/000131097. PMID 18453777
- [Background] Chisari G, Chisari EM, Francaviglia A, Chisari CG. The mixture of bifidobacterium associated with fructo-oligosaccharides reduces the damage of the ocular surface. Clin Ter. 2017 May-Jun;168(3):e181-e185. doi: 10.7417/T.2017.2002. PMID 28612893